CLINICAL TRIAL: NCT06529627
Title: Effect of Growth Differentiation Factor - 8 (GDF-8) on Pregnancy Rates in GnRH-agonist ICSI Cycles: A Prospective Cohort Study
Brief Title: GDF-8 Levels in ICSI Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mervat Sheikhelarab Elsedeek Ibrahim Omran, Professor of Obstetrics and Gynaecology, University of Alexandria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0107574
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Single group of infertile couple undergoing ICSI-ET with the standard long GnRH agonist protocol
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Long agonist protocol - ICSI-ET (Active Comparator)
  Interventions: Procedure: Long Gn-RH agonist protocol - Intracytoplasmic Sperm Injection

INTERVENTIONS:
Procedure: Long Gn-RH agonist protocol - Intracytoplasmic Sperm Injection — pituitary downregulation with GnRH agonist - ovarian stimulation with exogenous gonadotropin - hCG adminstration as trigger of oocyte maturation Oocyte retriveal via transvaginal ultrasound guided aspiration embryo transfer progesterone as luteal phase support

SUMMARY:
The aim of this study is to investigate the role of GDF-8 in regulating progesterone levels during controlled ovarian stimulation in patients undergoing ICSI-ET and to evaluate its effects on pregnancy rates.

The main questions are

* Does serum GDF-8 correlate with serum Progesterone levels during ovarian stimulation?
* Does serum GDF-8 serum level at different time-points during ovarian stimulation correlate with pregnancy rate?

participants will undergo ICSI-ET cycle using the long GnRH-agonist protocol and serum levels of GDF-8 and progesterone will be measured at three time-points during the trial: on day of hCG trigger administration, on day of oocyte pickup, and 14 days after embryo transfer

ELIGIBILITY:
Inclusion Criteria:

* The study population included women who underwent their first ICSI-ET cycles due to male and/or tubal factors or unexplained infertility, aged 20-35 years, whose BMI ranged from 19-29.9 kg/m2, with regular menstrual cycles

Exclusion Criteria:

* women with PCOS, couples with azoospermic husbands, women with poor ovarian reserve testing (AMH < 1.2 ng/dl and/or AFC < 5), women diagnosed with endometriosis, and women with medical comorbidities such as thyroid disorders, DM, hyperprolactinemia, etc.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 5 weeks after embryo transfer
  visualization of intra-uterine gestational sac with a pulsating fetal pole within 5 weeks of embryo transfer
Serum Growth Differentiation Factor - 8 (GDF-8) | three time-points: on day of trigger, on day of OPU, and 14 days after ET
  serum levels of GDF-8

CONTACTS AND LOCATIONS:
Locations (1):
- Shatby maternity university hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No